CLINICAL TRIAL: NCT04918836
Title: Immunological Markers Predictive of Response and Toxicity to Checkpoint in Metastatic Non-Small-cell Lung Cancers
Brief Title: Immunological Markers Predictive of Response and Toxicity to Checkpoint Inhibitors in Non-small Cell Lung Cancer
Acronym: IMMUNO-PREDICT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: Immuno-PREDICT ( 29BRC21.0021)
Record Dates: First submitted 2021-05-27; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective, observational, single-center study to determine the proportion of patients who have or will develop changes in biological markers of immunity during immunotherapy treatment.

DETAILED DESCRIPTION:
The study will run for 12 months with a 6-month follow-up at the inclusion of the last patient.

Patients will be included from the initiation of immunotherapy treatment regardless of the line.The routine immunological workup will be performed before the first immunotherapy infusion in order to analyze a certain number of immunological markers (autoantibodies, RF, LDH, complement (C3 C4), anti-tissue antibodies, lymphocyte immunophenotyping). This assessment will then be performed at progression, at the appearance of side effects requiring the immunotherapy to be stopped, or at 6 months of follow-up in case of continuation of the immunotherapy.

The investigators will evaluate the response to the treatment, the progression via re-evaluation assessments performed in standard practice (every 3 to 4 courses depending on the type of immunotherapy) as well as the appearance of side effects throughout the follow-up will be evaluate.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Metastatic non-small cell lung cancer
* Initiation of anti PDL1 therapy (NIVOLUMAB, PEMBROLIZUMAB or ATEZOLIZUAMB) in daily practice
* No objection made

Exclusion Criteria:

* Autoimmune disease diagnosed prior to initiation of immune checkpoint inhibitor therapy.
* Previous immune-modulating therapy (including corticosteroid therapy greater than 10 mg/day)
* Patient with prior checkpoint inhibitor therapy
* Patient with a contraindication to immunotherapy
* Patient under legal protection
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic non-small cell lung cancer receiving immunotherapy (NIVOLUMAB, PEMBROLIZUMAB or ATEZOLIZUMAB) regardless of the line of treatment in daily practice
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2021-10-08 (Estimated); Study Completion 2022-10-08 (Estimated)

PRIMARY OUTCOMES:
Change of biological markers of immunity under immunotherapy at 6 months | Day 0 and month 6 (M6)
  Determine the proportion of patients who have or will develop a change in biological markers of immunity under immunotherapy at 6 months or, failing that, at the end of the immunotherapy (FAN and/or RF and/or anti-tissue and/or decrease in acquired complement verified on the difference between 6 months and inclusion, lymphocyte immunophenotyping)

SECONDARY OUTCOMES:
Impact on Overall Survival (OS) and Progression Free Survival (PFS) | Day 0 and Six month after (M6)
  Determine if the presence of biological markers of autoimmunity at initiation or during anti-PD1/PDL1 immunotherapy influences overall survival or progression-free survival.
Impact on autoimmune toxicity | Day 0 and month 6 (M6)
  Determine if the presence of biological markers of autoimmunity (at inclusion, at 6 months or at progression) is associated with autoimmune toxicity (any clinical or biological autoimmune event regardless of its grade).
  Determine if the presence of biological markers of autoimmunity (at inclusion, at 6 months or at progression) is associated with autoimmune toxicity (any clinical or biological autoimmune event regardless of its grade).
Impact of complement | Day 0 and month 6 (M6)
  Determine if the decrease in complement at 6 months is associated with autoimmune toxicity.
Impact of autoimmune toxicity on OS | Day 0 and month 6 (M6)
  Determine if the occurrence of autoimmune toxicity during anti-PD1/PDL1 immunotherapy for non-small cell lung cancer influences the patient's overall survival.
Impact of autoimmune toxicity on PFS | Day 0 and month 6 (M6)
  Determine if the occurrence of autoimmune toxicity during anti-PD1/PDL1 immunotherapy for non-small cell lung cancer influences the patient's progression-free survival.
Impact of clinical factors | Day 0 and month 6 (M6)
  Determine if clinical factors (undernutrition, tumor mass, general condition) at initiation or during anti-PD1/PDL1 immunotherapy influence patient's overall survival and progression-free survival
Study the clinical factors influencing the immune profile | Day 0 and month 6 (M6)
  Study the clinical factors influencing the immune profile
Impact of CRP and lymphopenia | Day 0 and month 6 (M6)
  Determine if CRP and the presence of initial lymphopenia influence the presence or induction of an immunological abnormality

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 18 months and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.